CLINICAL TRIAL: NCT06185296
Title: The Intelligent Diabetes TelemonitoRing Using Decision Support to Treat Patients on Insulin Trial: Study Protocol for a Randomized Controlled Trial
Brief Title: The Intelligent Diabetes TelemonitoRing Using Decision Support to Treat Patients on Insulin Therapy
Acronym: DiaTRUST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry); DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Peter Vestergaard, MD, professor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DiaTRUST
Record Dates: First submitted 2023-12-06; First posted 2023-12-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Diabetes; Insulin; Telemedicine; Telehealth; Telemonitoring; CGM; Wearable devices; Adherence; Decision support; Algorithms
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intelligent telemonitoring (Experimental): The subjects will be telemonitored using the intelligent telemonitoring system. All subjects will use a CGM, a Fitbit, and a smart pen during the trial period. Staff at the endocrinology clinic will monitor the data and contact the subjects continuously throughout the trial (depending on the individual needs of each subject) using the intelligent telemonitoring system with embedded decision support to facilitate treatment evaluation and adjustments. The subjects will have access to a smartphone app that is able to provide a risk for nocturnal hypoglycemia before bed.
  Interventions: Device: Intelligent telemonitoring
- Telemonitoring (Active Comparator): The subjects will be telemonitored. All subjects will use a CGM, a Fitbit, and a smart pen during the entire trial period. Staff at the endocrinology clinic will monitor the data and contact the subjects continuously throughout the trial (depending on the individual needs of each subject)
  Interventions: Device: Telemonitoring
- Usual care (No Intervention): The subjects will wear a blinded CGM the first 20 days after inclusion, 20 days before the second visit to the trial site, and the final 20 days of the trial. The subjects will use a blinded smart pen throughout the trial period. Hence, the subjects cannot see their measured data during the trial and will not be monitored.

INTERVENTIONS:
Device: Intelligent telemonitoring — Telemonitoring using CGM, insulin pen data, and Fitbit data supported by data-driven decision support.
  Arms: Intelligent telemonitoring
Device: Telemonitoring — Telemonitoring using CGM, insulin pen data, and Fitbit data
  Arms: Telemonitoring

SUMMARY:
The trial is an open-label, randomized controlled trial. Patients with T2D on insulin therapy will be randomized to an intelligent telemonitoring group (intervention), a telemonitoring group (control), and a usual care group (control). Both the intelligent telemonitoring group and the telemonitoring group will use various devices at home. Hospital staff will monitor their data for three months. In the intelligent telemonitoring group, hospital staff and participants will be supported by decision-support algorithms in the management of insulin treatment.

DETAILED DESCRIPTION:
The DiaTRUST trial is an open-label randomized controlled trial with a three-month trial period. The trial will be conducted at Steno Diabetes Center North Jutland. Patients with T2D on insulin therapy will be randomized (3:1:1) to an intelligent telemonitoring group (intervention), telemonitoring alone (control), or a usual care group (control). Both telemonitoring groups will use an insulin pen, an activity tracker, a CGM, and a smartphone application throughout the trial period. Hospital staff (lab technicians and nurses) will monitor the telemonitoring groups' data and contact the subjects by telephone repeatedly throughout the trial period. For patients assigned to the intelligent telemonitoring group, decision support algorithms will provide hospital staff with insight and data overviews to support treatment evaluation and adjustment throughout the trial. Furthermore, patients in the intelligent telemonitoring group will have access to algorithms through a smartphone application that can provide a risk assessment before bed of nocturnal hypoglycemia. The usual care group will use a blinded CGM for the first 20 days after inclusion, 20 days before the second visit to the trial site, and 20 days before the end of trial and will use a blinded insulin pen for the entire period. The usual care groups' data will not be monitored during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years.
* Diagnosis of T2D for at least 12 months prior to the day of screening.
* Patients who are being treated with insulin or about to start insulin treatment (insulin naïve) willing to travel to trial site in North Denmark to attend in-person visits.
* Have internet at home, have MitID, and willingness to use a smartphone and the other devices used in the trial
* Signed informed consent.
* Ability to understand and read Danish.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Major surgery is planned during the trial period.
* Cancer diagnosis within five years prior to inclusion.
* Participation in other interventional trials.
* Limited literacy affecting the use of trial devices.
* Patient who has worn a CGM monitor less than 6 months prior to the trial.
* Terms that, in the opinion of the sub-investigator or investigator, render the participant unfit to conduct the trial, including lack of understanding of the trial or lack of physical or cognitive ability to participate.
* Patients treated with mixed insulin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
CGM time in range | At baseline to three months after randomization
  Change in CGM time in range (3,9-10,0 mmol/L)

SECONDARY OUTCOMES:
Concentration of HbA1c | At baseline to three months after randomization
  Change in HbA1c
CGM time in level 1 hypoglycemia (3.0-3.8 mmol/L) | At baseline to three months after randomization
  Change in CGM time in level 1 hypoglycemia (3.0-3.8 mmol/L)
CGM time in level 2 hypoglycemia (<3.0 mmol/L) | At baseline to three months after randomization
  Change in CGM time in level 2 hypoglycemia (<3.0 mmol/L)
CGM time in level 1 hyperglycemia (10.1-13.9 mmol/L) | At baseline to three months after randomization
  Change in CGM time above range (10.1-13.9 mmol/L)
CGM time in level 2 hyperglycemia (>13.9 mmol/L) | At baseline to three months after randomization
  Change in CGM time above range (>13.9 mmol/L)
Total daily units of insulin | At baseline to three months after randomization
  Change in total daily dose of insulin (units)
Number of hypoglycemic episodes | At baseline to three months after randomization
  Change in number of hypoglycemic episodes
Number of hyperglycemic episodes | At baseline to three months after randomization
  Change in number of hyperglycemic episodes
Body weight | At baseline to three months after randomization
  Change in body weight
Use of the telemonitoring equipment | Through study completion, an average of three months
  The frequency of use of the telemonitoring equipment
Time-to-target | At baseline to three months after randomization
  time until individualized treatment targets are reached
Time efficiency | At baseline to three months after randomization
  Between-group difference in time spent on contact with subjects and on treatment evaluation and adjustment by hospital staff
Fear of hypoglycemia | At baseline to three months after randomization
  Change in fear of hypoglycemia measured by Hypoglycemia Fear Survey-II short form (HFS-II short form) ranges from "never" to "almost always"
Diabetes-related quality of life | From baseline to three months after randomization
  Diabetes-related quality of life measured by the DIDP Questionnaire. Ranges from "very negative" to "very positive"
Health-related quality of life | From baseline to three months after randomization
  Health-related quality of life measured by the European Quality of Life Five Dimension Questionnaire (EQ-5D-5L). Options are not numeric in the descriptive part and follow the VAS scale in the second rating part ranging from 0 (The worst health you can image) to 100 (The best health you can image).
Change in patient adherence | From baseline to three months after randomization
  Patient adherence measured by the Insulin Adherence Questionnaire. Options are not numeric
Satisfaction with telemonitoring solution | At the three month assessment
  Satisfaction with telemonitoring solution measured by Digital Health Solution Satisfaction questionnaire (DHSS)
Change in treatment satisfaction | From baseline to three months after randomization
  Treatment satisfaction measured by the Diabetes Treatment Satisfaction Questionnaire (DTSQ)
Change in perceived competence in Diabetes | From baseline to three months after randomization
  Perceived competence in Diabetes measured by the Perceived competence in Diabetes questionnaire (PCD)
Change in CGM | Three months after randomization
  Change from baseline in CGM time in level 2 hypoglycemia (<3.0 mmol/L)

OTHER OUTCOMES:
Self-reported adherence | Through study completion, an average of 6 months
  Self-reported adherence insights from contacts between hospital staff and patients during the trial in the telemonitoring groups. Topics of conversation related to self-reported adherence will be collected based on predefined themes (e.g., missing basal dose due to forgetfulness, varying basal insulin dose during a week due to error on smartpen).
Insulin doses | Through study completion, an average of 6 months
  Any differences in the use of insulin in terms of dosing between the three groups are examined based on data from the insulin pens, e.g., differences in the amount of insulin taken per patient (measured by units per insulin type), and differences in change in insulin dose during the trial period (measured by units).
Insulin dosing time | Through study completion, an average of 6 months
  Any differences in the use of insulin in terms of timing of the dosing between the three groups are examined based on data from the insulin pens, e.g., differences in injection patterns.
Number of CGM days worn | During the intervention and active comparator
  Number of days that the subjects wear the CGM
CGM percentage of time active | During the intervention and active comparator
  Percentage of time that the CGM is active
Mean glucose | At baseline to three months after randomization
  Mean glucose levels (mmol/l) measured by CGM
Glycemic variability | At baseline to three months after randomization
  Glycemic variability - percentage of coefficient of variation
Glucose management indicator | At baseline to three months after randomization
  Change in estimated A1c (%) derived from CGM
Dietary habits | At baseline to three months after randomization
  Change in diet habits collected by predefined questions. Options are not numeric.
Exercise habits | At baseline to three months after randomization
  Change in exercise habits collected by predefined questions. Options are not numeric.
Self-reported information on diet and exercise habits | Through study completion, an average of 3 months
  Self-reported information on diet and exercise habits collected from the contacts between hospital staff and patients throughout the trial period. Notes will be collected based on these conservations on e.g., the patient's realising impact of certain foods in blood glucose variations, patient and hospital staff agree to try reach a higher number of steps per day.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vestergaard, MD, PhD, Principal Investigator — Steno Diabetes Center North Denmark
Locations (1):
- Department of Endocrinology, Aalborg, North Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomsen CHN, Norlev JTD, Hangaard S, Jensen MH, Hejlesen O, Cohen SR, Kofoed-Enevoldsen A, Kristensen SNS, Aradottir TB, Kaas A, Vestergaard P, Kronborg T. The intelligent diabetes telemonitoring using decision support to treat patients on insulin therapy (DiaTRUST) trial: study protocol for a randomized controlled trial. Trials. 2024 Nov 8;25(1):744. doi: 10.1186/s13063-024-08588-7. PMID 39511648